CLINICAL TRIAL: NCT06985498
Title: Safety and Efficacy of CD22/CD19 CAR-T and Blinatumomab Combined With Auto-HSCT Sandwich Strategy as Consolidation Therapy for B-cell Acute Lymphoblastic Leukemia
Brief Title: CD22/CD19 CAR-T and Blinatumomab Combined With Auto-HSCT Sandwich Strategy as Consolidation Therapy for B-ALL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Prof., The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZCART03
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphobkastic Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sandwich strategy (Experimental)
  Interventions: Combination Product: Sandwich stratergy

INTERVENTIONS:
Combination Product: Sandwich stratergy — The patients received blinatumoab after standard induction and consolidation chemotherapy. Autologous stem cells mobilization and collection were performed after blinatumomab. Auto-HSCT was proceeded after successful stem cell collection. CD22 and CD19 CAR-T cells were re-infused 2 days after stem cell reinfusion.

SUMMARY:
Chimeric antigen receptor T-cell (CAR-T) therapy has achieved remarkable efficacy in B-cell acute lymphoblastic leukemia (B-ALL). However, relapse after CAR-T has been a major issue. Multi-antigen CAR T and combination with other regimens may reduce the relapse rate. We conducted CD22/CD19 CAR T-cells and blinatumoab combined with auto-HSCT "sandwich " strategy as consolidation therapy in patients with B-ALL. The main Purpose of this study was to observe the safety and efficacy of this new strategy.

ELIGIBILITY:
Inclusion Criteria:

1. subjects with a primary diagnosis of B-ALL who have any of the following: (a) no suitable allogeneic HSCT donor. (b) refusal of allogeneic HSCT;
2. positive expression of CD19 and CD22 in peripheral blood or bone marrow primary cells detected by flow cytometry;
3. cardiac ultrasound left ventricular ejection fraction ≥ 50%; Creatinine ≤ 1.6 mg/dl; alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the normal range and total bilirubin ≤ 2.0 mg/dl; Pulmonary function ≤ grade 1 dyspnea (CTCAE v5.0) with oxygen saturation > 91% without oxygenation;
4. subjects aged 15-65 years (including 15 and 65 years), regardless of gender;
5. T-cell amplification test pass;
6. expected survival > 3 months.

Exclusion Criteria:

1. patients with recurrence of only isolated extramedullary lesions;
2. combination of other malignant tumors;
3. previously treated with anti-CD19 or/and CD22 or/and CD3 therapies;
4. immunosuppressants use within 2 weeks prior to signing informed consent or plan to immunosuppressants after signing informed consent;
5. uncontrolled active infections;
6. HIV infection;
7. active hepatitis B or hepatitis C infection;
8. history of severe tachyphylaxis to aminoglycoside antibiotics;
9. history or presence of clinically relevant Central Nervous System (CNS) pathology, such as epilepsy, generalized seizure disorder, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive

SECONDARY OUTCOMES:
leukemia free survival | 2 years
  It is measured from the date of achievement of a remission after blinatumomab until the date of relapse from CR, or CRi, or death from any cause; patients not known to have any of these events are censored on the date they were last examined.
Number of adverse events | 2 years
  Adverse events are evaluated with CTCAE V5.0 among Sandwich stratergy.